CLINICAL TRIAL: NCT03217695
Title: A Pilot Study on the Effect of Mindfulness-based Yoga on Youth With Persistent Concussion Symptoms: Bridging Neurophysiological and Functional Outcomes
Brief Title: A Study on the Effect of Mindfulness-based Yoga on Youth With Persistent Concussion Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BloorviewKR_MBY
Record Dates: First submitted 2017-06-19; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-06

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury
Keywords: Heart rate variability; Self-efficacy; Pediatrics; Mindfulness-based yoga; Symptoms
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-based Yoga Arm (Experimental): 8-week period, 1x/week for 45-60 minutes/session. Sessions 1-2: Participants instructed to focus their attention on their breath, and the physical sensations in their bodies while holding the yoga postures, to develop sustained and focused attention. Sessions 3-4: exploring the sensorial qualities of physical sensation in the body whether pleasant or unpleasant and to notice thoughts and label them (e.g., "planning", "remembering"), and to the same with emotions (e.g., "worry", "frustration", "fear") to practice disengaging from automatic associative thinking. Session 6-8: Instructor will guide participants to allow sensations of discomfort or effort to be as they are and to bring awareness to automatic patterns of reactivity. The goal is to foster distress tolerance, provide opportunities for participants to practice self-care, and allow an opportunity to observe and respond skillfully, instead of react automatically, to unpleasant stimuli (sensations, emotions).
  Interventions: Behavioral: Mindfulness-based Yoga Arm

INTERVENTIONS:
Behavioral: Mindfulness-based Yoga Arm

SUMMARY:
Mild traumatic brain injury (mTBI), also known as concussion, is of great concern in the youth population, with incidences of injury steadily increasing within the past few years. Current Canadian estimates have indicated that the total rate of concussions per 100,000 increased from 467 to 754 for boys and from 209 to 441 for girls from 2003-2010. As defined by the recent Zurich Consensus statement, concussion is a pathophysiological injury induced by biomechanical forces, which can be caused by impact to the head, neck or body. In 10-20% of youth, concussion symptoms persist in the weeks, months or even years following the injury. Consequently, youth with persistent concussion symptoms are unable to fully participate in the meaningful activities (e.g. attending school, engaging with friends and community) they did prior to the injury and experience a reduced quality of life.

Persistent concussion symptoms in youth requires an approach that directly addresses the rumination and attention to distressful thoughts about their functional performance, while still promoting appropriate levels of physical and cognitive demands. Targeting these constructs may shift the focus away from symptoms, while building self-efficacy and enhancing participation in daily activities. Mindfulness-based yoga (MBY) is a mind-body intervention that uses physical yoga poses, purposeful breathing techniques and a focus on being in the present moment. MBY encourages participants to develop moment-to-moment awareness of physical sensations, emotions, and thoughts, and promotes the cultivation of non-judgemental and accepting relationships to personal experiences. In chronic pain, fibromyalgia, mental health and now TBI populations, MBY has demonstrated benefits in physical (i.e. increased muscle strength, endurance), psychological (i.e. decreased stress, increased self-efficacy), cognitive (i.e. increased concentration) and social (i.e. emotional regulation, improved mood) domains. Although mindfulness based yoga has been validated as a form of rehabilitation in the adult population, its applicability for youth with persistent concussion symptoms has yet to be explored. Understanding the impact of a MBY intervention on this population may enhance management of persistent symptoms and ultimately, participation in meaningful activities.

In addition to the functional sequelae that ensue following this injury, concussion in both the acute and persistent phases is being recognized as a neurophysiological injury. Traditional methods of assessment following concussion place emphasis on subjective self-report and administration of neuropsychological batteries. These assessments are used in an effort to return the youth to activity (i.e school, sport). However, these methods can be unreliable as youth have a high incentive to return to play and neurocognitive resolution does not necessarily equate to pre-injury function. To augment these measures, an objective indicator of neurophysiological stress is needed. Heart rate variability (HRV) is an objective, neurophysiological indicator of autonomic nervous system functioning. HRV is quantified by measuring the time intervals between heartbeats. Increased variability in heart rate (i.e. increased HRV) is seen as healthy neurophysiological function, demonstrating an individual's ability to adapt and be flexible to the demands of the environment. Conversely, decreased HRV is demonstrative of an individual's reduced ability to respond flexibly to their environment. Investigating the impact of persistent concussion symptoms on HRV has the potential to enhance our understanding of autonomic nervous system functioning in the chronic phases of this injury for an understudied population.

The specific objectives are to: (1) adapt the MBY intervention protocol to suit the unique needs of youth with mTBI (i.e. safety, fatigue), (2) collect data on the impact of MBY on HRV, self-efficacy and participation, (3) describe changes in HRV, self-efficacy and participation associated with MBY across pre-intervention, post-intervention and 3 months following intervention, (4) identify if post concussion symptoms change (i.e. increase or decrease) following MBY and (5) identify if changes in post concussion symptoms occur with changes in HRV, self-efficacy and participation.

ELIGIBILITY:
Inclusion Criteria:

* Youth between 13-18 years old;
* Persistent concussion symptoms greater than 1 month.

Exclusion Criteria:

* Less than 13 years old or greater than 18 years old;
* Non-English speaking;
* Severe (unmanaged) psychiatric diagnosis;
* Neurological disease;
* Diagnosed cardiac issues.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Change in Children's Assessment of Participation and Employment (CAPE) from pre-intervention to 3 month follow-up | Pre-intervention, post-intervention (within 1 week following 8-week intervention), 3 month follow-up
  Participants are asked to complete the 55-item questionnaire and answer questions about an activity based on five dimensions of participation: diversity (number of activities done), intensity, (with whom the youth does an activity with), where (they do it) and enjoyment of activities (King et al., 2007).
Change in Self-Efficacy Questionnaire for Children (SEQ-C) from pre-intervention to 3 month follow-up | Pre-intervention, post-intervention (within 1 week following 8-week intervention), 3 month follow-up
  Participants are asked to rate their perceived ability to accomplish a task between 1 (not at all) to 5 (very well). The questions cover three domains of self-efficacy, namely social, academic and emotional.
Change in Heart rate variability from pre-intervention to 3 month follow-up | Pre-intervention, during each of the 8 weeks of mindfulness-based yoga (for 24 hours starting at 6PM when each of the yoga sessions begins until 6PM the following day), post-intervention (within 1 week following 8-week intervention), 3 month follow-up
  Time (seconds) of beat-to-beat intervals, measured over a 24 hour recording

SECONDARY OUTCOMES:
Post-Concussion Symptom Inventory (PCSI) | Pre-intervention, post-intervention (within 1 week following 8-week intervention), 3 month follow-up
  It is a 21-item self-report measure where symptom severity is rated on a scale of 0 to 6 (0= not at all, 3= moderate, 6=severe) for symptoms that occur within physical, cognitive, fatigue and emotional domains
Godin Leisure-Time Exercise Questionnaire (GLTE) | Pre-intervention, post-intervention (within 1 week following 8-week intervention), 3 month follow-up
  It is a self-report measure that assesses weekly physical activity engagement by asking participants to indicate how many times per week they engage in strenuous (heart beats rapidly), moderate (not exhausting) or mild exercise (minimal effort).

CONTACTS AND LOCATIONS:
Overall Officials: Nick Reed, MScOT, PhD, Principal Investigator — Bloorview Research Institute, Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hopsital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Abaji JP, Curnier D, Moore RD, Ellemberg D. Persisting Effects of Concussion on Heart Rate Variability during Physical Exertion. J Neurotrauma. 2016 May 1;33(9):811-7. doi: 10.1089/neu.2015.3989. Epub 2015 Oct 8. PMID 26159461
- [Background] Azulay J, Smart CM, Mott T, Cicerone KD. A pilot study examining the effect of mindfulness-based stress reduction on symptoms of chronic mild traumatic brain injury/postconcussive syndrome. J Head Trauma Rehabil. 2013 Jul-Aug;28(4):323-31. doi: 10.1097/HTR.0b013e318250ebda. PMID 22688212
- [Background] Belanger HG, Kretzmer T, Vanderploeg RD, French LM. Symptom complaints following combat-related traumatic brain injury: relationship to traumatic brain injury severity and posttraumatic stress disorder. J Int Neuropsychol Soc. 2010 Jan;16(1):194-9. doi: 10.1017/S1355617709990841. Epub 2009 Sep 17. PMID 19758488
- [Background] Blechert J, Michael T, Grossman P, Lajtman M, Wilhelm FH. Autonomic and respiratory characteristics of posttraumatic stress disorder and panic disorder. Psychosom Med. 2007 Dec;69(9):935-43. doi: 10.1097/PSY.0b013e31815a8f6b. Epub 2007 Nov 8. PMID 17991823
- [Background] Conder RL, Conder AA. Heart rate variability interventions for concussion and rehabilitation. Front Psychol. 2014 Aug 13;5:890. doi: 10.3389/fpsyg.2014.00890. eCollection 2014. PMID 25165461
- [Background] Deshpande S, Nagendra HR, Nagarathna R. A randomized control trial of the effect of yoga on Gunas (personality) and Self esteem in normal healthy volunteers. Int J Yoga. 2009 Jan;2(1):13-21. doi: 10.4103/0973-6131.43287. PMID 21234210
- [Background] Galantino ML, Galbavy R, Quinn L. Therapeutic effects of yoga for children: a systematic review of the literature. Pediatr Phys Ther. 2008 Spring;20(1):66-80. doi: 10.1097/PEP.0b013e31815f1208. PMID 18300936
- [Background] Hofmann SG, Sawyer AT, Witt AA, Oh D. The effect of mindfulness-based therapy on anxiety and depression: A meta-analytic review. J Consult Clin Psychol. 2010 Apr;78(2):169-83. doi: 10.1037/a0018555. PMID 20350028
- [Background] Jonsson C, Andersson EE. Mild traumatic brain injury: a description of how children and youths between 16 and 18 years of age perform leisure activities after 1 year. Dev Neurorehabil. 2013;16(1):1-8. doi: 10.3109/17518423.2012.704955. Epub 2012 Oct 3. PMID 23030702
- [Background] King GA, Law M, King S, Hurley P, Hanna S, Kertoy M, Rosenbaum P. Measuring children's participation in recreation and leisure activities: construct validation of the CAPE and PAC. Child Care Health Dev. 2007 Jan;33(1):28-39. doi: 10.1111/j.1365-2214.2006.00613.x. PMID 17181750
- [Background] Leddy JJ, Kozlowski K, Fung M, Pendergast DR, Willer B. Regulatory and autoregulatory physiological dysfunction as a primary characteristic of post concussion syndrome: implications for treatment. NeuroRehabilitation. 2007;22(3):199-205. PMID 17917170
- [Background] Macpherson A, Fridman L, Scolnik M, Corallo A, Guttmann A. A population-based study of paediatric emergency department and office visits for concussions from 2003 to 2010. Paediatr Child Health. 2014 Dec;19(10):543-6. doi: 10.1093/pch/19.10.543. PMID 25587234
- [Background] McCrory P, Meeuwisse W, Aubry M, Cantu B, Dvorak J, Echemendia R, Engebretsen L, Johnston K, Kutcher J, Raftery M, Sills A, Benson B, Davis G, Ellenbogen R, Guskiewicz K, Herring SA, Iverson G, Jordan B, Kissick J, McCrea M, McIntosh A, Maddocks D, Makdissi M, Purcell L, Putukian M, Schneider K, Tator C, Turner M. Consensus statement on Concussion in Sport - The 4th International Conference on Concussion in Sport held in Zurich, November 2012. Phys Ther Sport. 2013 May;14(2):e1-e13. doi: 10.1016/j.ptsp.2013.03.002. No abstract available. PMID 23664041
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Reed N, Murphy J, Dick T, Mah K, Paniccia M, Verweel L, Dobney D, Keightley M. A multi-modal approach to assessing recovery in youth athletes following concussion. J Vis Exp. 2014 Sep 25;(91):51892. doi: 10.3791/51892. PMID 25285728
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Zemek RL, Farion KJ, Sampson M, McGahern C. Prognosticators of persistent symptoms following pediatric concussion: a systematic review. JAMA Pediatr. 2013 Mar 1;167(3):259-65. doi: 10.1001/2013.jamapediatrics.216. PMID 23303474